CLINICAL TRIAL: NCT00093925
Title: Evaluation of Clevidipine in the Postoperative Treatment of Hypertension Assessing Safety Events (With Nicardipine as Active Comparator) (ECLIPSE-NIC)
Brief Title: Clevidipine in the Postoperative Treatment of Hypertension (ECLIPSE-NIC)
Acronym: ECLIPSE-NIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC-CLV-03-05; ECLIPSE-NIC (Other: Sponsor)
Record Dates: First submitted 2004-10-07; First posted 2004-10-08 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: Postoperative hypertension
MeSH Terms: conditions — Hypertension | interventions — clevidipine; Nicardipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clevidipine (Experimental): Clevidipine (0.5 mg/mL in 20% lipid emulsion) was initiated after insertion of an arterial line upon the occurrence of postoperative hypertension, as determined by the investigator, and was administered intravenously (IV) at an initial infusion rate of 0.4 μg/kg/min (non weight-based equivalent is 2 mg/h). Clevidipine was titrated to blood pressure lowering effect by doubling increments approximately every 90 seconds up to a maximum infusion rate of 3.2 μg/kg/min (16 mg/h). Infusion rates above 3.2 μg/kg/min were permitted up to the maximum infusion rate of 8.0 μg/kg/min. Treatment was maintained as long as was deemed clinically necessary or until discharge from the ICU. Infusion rates between 4.4 and 8.0 μg/kg/min were to be administered for no more than 2 hours.
  Interventions: Drug: clevidipine
- nicardipine (Active Comparator): Nicardipine (NIC) was initiated after insertion of an arterial line upon the occurrence of postoperative hypertension, as determined by the investigator, and was administered intravenously as per institutional practice. Treatment was maintained as long as was deemed clinically necessary or until discharge from the ICU.
  Interventions: Drug: nicardipine

INTERVENTIONS:
Drug: clevidipine
  Other Names: clevidipine, Cleviprex
  Arms: clevidipine
Drug: nicardipine
  Arms: nicardipine

SUMMARY:
The purpose of this study is to establish the safety of clevidipine in the treatment of postoperative hypertension. Approximately 250-500 patients with postoperative hypertension after undergoing coronary artery bypass grafting (CABG), off-pump coronary artery bypass (OPCAB) or minimally invasive direct coronary artery bypass (MIDCAB) surgery and/or valve replacement/repair procedures were anticipated to be randomly assigned to one of two treatment groups: clevidipine or nicardipine.

DETAILED DESCRIPTION:
The primary objective was to establish the safety of clevidipine in the treatment of postoperative hypertension, as assessed by comparing the incidences of death, stroke, MI and renal dysfunction in the clevidipine and nicardipine treatment groups from the initiation of study drug infusion through postoperative Day 30. Secondary objectives were to evaluate the efficacy of study drug, assessed by the blood pressure (BP) lowering effect, and additional safety variables.

ELIGIBILITY:
Prerandomization Inclusion Criteria:

* Provide written informed consent before initiation of any study related procedures.
* Be at least 18 years of age
* Be scheduled for Coronary Artery Bypass Grafting (CABG), Off Pump Coronary Artery Bypass (OPCAB), Minimally Invasive Direct Coronary Artery Bypass (MIDCAB) surgery, and/or valve replacement/repair surgery

Prerandomization Exclusion Criteria:

* Women of child-bearing potential (unless they have a negative pregnancy test)
* Recent cerebrovascular accident (within 3 months before randomization)
* Known intolerance to calcium channel blockers
* Known or suspected hypersensitivity to nicardipine
* Allergy to soybean oil or egg lecithin (components of the lipid vehicle)
* Pre-existing permanent ventricular pacing
* Any other disease or condition, which, in the judgment of the investigator would place a patient at undue risk by being enrolled in the trial
* Participation in another therapeutic drug or therapeutic device trial within 30 days of starting study

Postrandomization Inclusion Criteria:

* Expected to survive beyond 24 hours post-surgical procedure
* No surgical complications or conditions, present or anticipated, that preclude them from inclusion in the study
* Determined to be hypertensive postoperatively as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2004-05; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Incidence of death, stroke, MI, and renal dysfunction | Initiation of study drug infusion through post-operative Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Lloyd, MD, Study Director — The Medicines Company - Medical Director, Clinical Operations
Locations (9):
- United States (9):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Wesley Medical Center, Wichita, Kansas
  - Touro Infirmary, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Columbia University - College of Physicians and Surgeons, New York, New York
  - Jack D. Weller Hospital, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - VA Medical Center McGuire, Richmond, Virginia

REFERENCES:
- [Result] Aronson S, Dyke CM, Stierer KA, Levy JH, Cheung AT, Lumb PD, Kereiakes DJ, Newman MF. The ECLIPSE trials: comparative studies of clevidipine to nitroglycerin, sodium nitroprusside, and nicardipine for acute hypertension treatment in cardiac surgery patients. Anesth Analg. 2008 Oct;107(4):1110-21. doi: 10.1213/ane.0b013e31818240db. PMID 18806012